CLINICAL TRIAL: NCT04558671
Title: Bronchial REmodeling in Severe Preschool Wheezing chIldren and Risk of Exacerbation
Brief Title: Preschool Bronchial Remodeling and Risk of Exacerbation
Acronym: RESPIRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/32
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Preschool Severe Asthma
Keywords: exacerbation; children; asthma; bronchial remodeling; wheezing
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: asthma exacerbations — to collect the number of asthma exacerbations between the 2 latent classes of patients within the year following bronchoscopy

SUMMARY:
Bronchial remodeling is an abnormal tissue repair process of the bronchial wall components that characterizes severe asthma which can include epithelial abrasion, thickening of the reticular basement membrane (RBM), an increase in bronchial fibrosis, blood vessel count, mucosal gland mass and/or bronchial smooth muscle (BSM) mass. We identified using latent class analysis two classes of patients. Compared to the second class, the first class was characterized by an increase in RBM thickness, blood vessel count, BSM mass and a decrease in RBM-BSM distance, mucus gland mass and bronchial fibrosis. We then hypothesized that this first latent class identified children at risk of asthma exacerbations.

DETAILED DESCRIPTION:
Asthma is the most frequent chronic disease in children. Severe asthma is characterized by airway hyperresponsiveness, bronchial inflammation and bronchial remodeling 1. Bronchial remodeling is an abnormal tissue repair process of the bronchial wall components which can include epithelial abrasion, thickening of the reticular basement membrane (RBM), an increase in bronchial fibrosis, blood vessel count, mucosal gland mass and/or bronchial smooth muscle (BSM) mass. At preschool age (before 6 years old), asthmatic children constitute a heterogeneous population and several classifications have been proposed to identify distinct phenotypes according to the chronology of asthma 2, the triggers of asthma 3, the trajectory of lung function as measured by forced expiratory volume in 1 second (FEV1) 4 or according to a combination of clinical and inflammatory variables 5. More recently, we demonstrated for the first time using latent class analysis (LCA) that subgroups of severe asthmatic children could also be identified according to bronchial remodeling parameters (unpublished data). Indeed, we identified two latent classes of patients. Compared to the second class, the first latent class was characterized by an increase in RBM thickness, blood vessel count, BSM mass and a decrease in RBM-BSM distance, seromucosal gland mass and bronchial fibrosis (unpublished data). Since, previous studies showed that bronchial remodeling could have negative impact on the patients' outcomes, we therefore hypothesized that the latent classes identified from the bronchial remodeling data in severe preschool asthmatic children included in the "P'tit Asthme" study (NCT02806466) could identify children at risk of asthma exacerbations requiring systemic corticosteroids therapy.

ELIGIBILITY:
Inclusion Criteria:

* To have been previously included in the "P'tit Asthme" study (NCT02806466)
* To have performed bronchoscopy with analyzable biopsies
* To have been asthmatic at the inclusion in the P'tit Asthme study (NCT02806466)

Exclusion Criteria:

• To refuse the use of children data as expressed by representatives of parental authority

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Severe preschool wheezers (1-5 years old) according to ERS and ATS modified criteria and requiring flexible bronchoscopy according to ERS guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations | 1 year
  Number of asthma exacerbations requiring systemic corticosteroid therapy within the year following the bronchoscopy performed in the "P'tit Asthme" study.

SECONDARY OUTCOMES:
Presence of the exacerbation prone asthma | 1 year
  Presence of the exacerbation prone asthma defined by the occurrence of 3 or more asthma exacerbations requiring systemic corticosteroid therapy within one year
Number of asthma exacerbations requiring systemic corticosteroid therapy | 1 year
  Number of asthma exacerbations requiring systemic corticosteroid therapy each month within the year following the bronchoscopy performed in the P'tit Asthme study.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux, Aquitaine
  - CHU de Toulouse, Toulouse, Occitanie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayon M, Beaufils F, Esteves P, Campagnac M, Maurat E, Michelet M, Siao-Him-Fa V, Lavrand F, Simon G, Begueret H, Berger P; P'tit Asthme Study Group. Bronchial Remodeling-based Latent Class Analysis Predicts Exacerbations in Severe Preschool Wheezers. Am J Respir Crit Care Med. 2023 Feb 15;207(4):416-426. doi: 10.1164/rccm.202205-0913OC. PMID 36108144